CLINICAL TRIAL: NCT06821984
Title: Evaluation of Cyanoacrylate as an Alternative to Sutures in Free Gingival Graft Stabilization: Effects on Graft Shrinkage, Microcirculation, and Postoperative Healing
Brief Title: Evaluation of Cyanoacrylate as an Alternative to Sutures in Free Gingival Graft Stabilization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Zeynep Turgut Çankaya, Principal Investigator, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 84 / 12.08.2018
Record Dates: First submitted 2025-02-05; First posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Gingival Recession
MeSH Terms: conditions — Gingival Recession | interventions — Sutures

STUDY DESIGN:
Intervention Model Description: Parallel-group randomized controlled trial
  Two intervention groups:
  Suture group (control): FGG secured with conventional sutures. Cyanoacrylate group (test): FGG secured using cyanoacrylate tissue adhesive without sutures.
Who Masked: Participant, Outcomes Assessor
Masking Description: his study is designed as a randomized controlled clinical trial (RCT) to evaluate the efficacy of cyanoacrylate (CA)-based adhesive in stabilizing free gingival grafts (FGG) compared to traditional sutures. The study model includes the following key components:Standardized FGG procedure performed by the same experienced periodontist.
  Grafts harvested from the hard palate and adapted to the recipient site. Hemostasis at the donor site managed with either traditional methods (sutures) or cyanoacrylate.
  Graft stabilization: Sutures (control) vs. cyanoacrylate (test).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cyanoacrylate (test). (Experimental): FGG secured using cyanoacrylate tissue adhesive without sutures.
  Interventions: Procedure: FGG secured using cyanoacrylate tissue adhesive without sutures.
- Suture group (control) (No Intervention): GG secured with conventional sutures.

INTERVENTIONS:
Procedure: FGG secured using cyanoacrylate tissue adhesive without sutures. — The intervention involved securing the free gingival graft (FGG) using cyanoacrylate adhesive instead of conventional sutures. After harvesting the graft from the hard palate, hemostasis at the donor site was achieved with gauze compression. The recipient site was prepared with a partial-thickness dissection to ensure a stable graft bed. In the intervention group, cyanoacrylate adhesive was applied along the margins of the graft and underlying periosteal bed, ensuring complete coverage without the use of sutures. The adhesive polymerized within seconds, creating an immediate bond between the graft and recipient site, minimizing micro-movements and reducing the need for additional fixation.
  Arms: cyanoacrylate (test).

SUMMARY:
Free gingival graft (FGG) is a widely used periodontal plastic surgery technique for treating gingival recession, increasing keratinized gingiva width, and enhancing peri-implant soft tissues. Despite its predictable outcomes, donor site morbidity, postoperative pain, and graft contraction remain challenges.

This study evaluates the efficacy of cyanoacrylate for securing FGGs without sutures at the recipient site and accelerating donor site healing. Laser Doppler flowmetry (LDF) and digital measurement techniques were used to objectively assess microcirculation and graft shrinkage.

Although previous research has investigated dimensional changes and vascular dynamics in FGG healing, no study has assessed absolute area changes in cyanoacrylate-fixed grafts or its impact on microcirculation at both the donor and recipient sites.

This randomized controlled clinical trial compares cyanoacrylate and suture fixation in early healing, focusing on graft shrinkage, microcirculation, and postoperative pain. By analyzing the effects of cyanoacrylate on wound healing and blood flow, this study aims to optimize surgical outcomes and improve patient recovery.

DETAILED DESCRIPTION:
Free gingival graft (FGG) is a widely used periodontal plastic surgery technique for treating gingival recession, increasing keratinized gingiva width, and enhancing peri-implant soft tissues. This procedure helps improve oral hygiene by creating a keratinized tissue barrier that resists frictional forces. While FGG is considered the gold standard due to its predictable success, donor site healing remains a challenge, often associated with postoperative pain, bleeding, and discomfort.

FGG involves two wound sites: the recipient and the donor site. The donor site, typically the hard palate, heals by secondary intention. Research has focused on minimizing donor site morbidity by exploring various biomaterials, growth factors, and wound healing strategies, such as platelet-rich fibrin (PRF), laser therapy, and chemotherapeutic agents. Covering the donor site aims to reduce bacterial contamination, accelerate healing, and decrease pain. Recent advancements in biomaterials and tissue adhesives have been explored to optimize this process.

At the recipient site, graft adaptation and long-term stability are crucial for success. Proper vascularization, integration, and esthetic outcomes depend on biological responses and surgical techniques. Traditional suturing methods, while effective, contribute to graft contraction due to tissue trauma and increased hematoma formation. Alternative stabilization methods, such as fibrin glue, staples, adhesive tapes, and cyanoacrylate-based adhesives, have been explored to minimize these effects.

Cyanoacrylate (CA)-based adhesives are promising biomaterials for tissue fixation due to their high adhesion strength, rapid polymerization, and stability in moist environments. First introduced for FGG stabilization by Hoexter in 1978, CA adhesives have demonstrated bacteriostatic properties, slow biodegradability, and reduced postoperative pain compared to sutures. Butyl cyanoacrylate (BCA) adhesives, in particular, provide hemostatic effects and facilitate rapid wound closure, potentially reducing complications such as graft shrinkage and donor site bleeding.

Previous studies on FGG contraction assumed uniform linear shrinkage, which may not accurately reflect the actual healing process. Digital measurement techniques provide more precise assessments by accounting for the irregular surface morphology of healing grafts. Additionally, microcirculatory changes play a critical role in graft survival, with vascular connections forming by the third day and sinusoidal vascular loops developing by day five (Nobuto et al., 1988). Laser Doppler flowmetry (LDF) is a non-invasive tool used to evaluate blood flow dynamics in gingival wound healing, providing objective and repeatable microcirculatory data.

Despite existing research on FGG healing and donor site dynamics, no study has comprehensively assessed the absolute area changes of cyanoacrylate-secured grafts or its impact on microcirculation at both the donor and recipient sites. This randomized controlled clinical trial aims to compare suture fixation and cyanoacrylate tissue adhesives during early healing. Key parameters include graft shrinkage, microcirculation, and postoperative pain.

By integrating LDF and digital measurement techniques, this study seeks to provide objective data on the effects of cyanoacrylate on blood flow and tissue healing. The findings may contribute to optimizing surgical outcomes, improving patient comfort, and reducing complications associated with FGG procedures.

ELIGIBILITY:
Inclusion Criteria:

Presence of at least one site with <2 mm of keratinized tissue, diagnosed using the functional test (borderline between movable and immovable tissue) [36].

Limited to the lower central and lateral incisors, canines, and first and second premolars in each patient.

Exclusion Criteria:

Gingival thickness ≥1 mm. Absence of a pulling frenum in the keratinized tissue. No parafunctional habits. No history of mucogingival or periodontal surgery. No restorations or crown prostheses.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Graft Shrinkage Assessed via Digital Image Analysis | 1 month
  Graft shrinkage is measured digitally using image analysis software to assess dimensional stability over time. Standardized clinical photographs are taken at predefined time points, and changes in graft dimensions are quantified using calibrated digital measurement tools. Measurements include changes in graft surface area and linear contraction over the follow-up period.
Microcirculation dynamics | 1 week
  Assessed using laser Doppler flowmetry (LDF) at different time points postoperatively.

SECONDARY OUTCOMES:
Postoperative Pain Assessment Using the Visual Analog Scale (VAS) | 1 week
  Postoperative pain will be assessed using the Visual Analog Scale (VAS), a 10 cm linear scale ranging from 0 to 10. The minimum value (0) represents 'no pain,' while the maximum value (10) indicates 'worst imaginable pain.' Higher scores correspond to greater pain intensity, indicating a worse outcome.
Healing Assessment at Donor and Recipient Sites Using Clinical Parameters | 1 week
  Healing at donor and recipient sites will be evaluated using clinical parameters, including epithelialization, wound closure, and presence of inflammation. Healing will be assessed at predefined time points through standardized clinical examination by a calibrated periodontist. Each parameter will be graded using Gingival Indices (0-3), where 0 indicates no healing/inflammation and 3 represents complete healing/no inflammation. Higher scores indicate better healing outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Turgut Çankaya, Ass Prof, Principal Investigator — Gazi University
Locations (1):
- Gazi University Faculty of Dentistry Department of Periodontology, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Upon Request
Supporting Information: Study Protocol, ICF, CSR
Time Frame: during the publishing
Access Criteria: upon request with principal investigator